CLINICAL TRIAL: NCT06131593
Title: TAP Block With Dexamethasone Versus TAP Block With Methyl-prednisolone as a Pain Treatment Modality After Total Abdominal Hysterectomy Procedures: Randomized Controlled Trial
Brief Title: TAP Block With Methyl-prednisolone as a Pain Treatment Modality After Total Abdominal Hysterectomy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-139-2023
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Local Anesthetic; Ultrasound; Pain, Acute
Keywords: ultrasound; TAP block; Hystrectomy; methyl prednisolone
MeSH Terms: conditions — Acute Pain | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane; Dexamethasone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Patients will be divided in to two groups; TAPB with dexamethasone as an adjuvant to local anesthetic Gr A(n=25) and TAPB with methyl prednisolone as an adjuvant to local anesthetic Gr B(n=25).
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and assessing study outcomes will be blinded to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TAPB-D (n=25) (Experimental): Patients in this group will receive TAPB with dexamethasone as an adjuvant to local anesthetic.
  Interventions: Drug: TAPB with dexamethasone as an adjuvant to local anesthetics
- Group TAPB-M (n=25) (Active Comparator): Patients in this group will receive TAPB with methylprednisolone as an adjuvant to local anesthetic.
  Interventions: Drug: TAPB with methylprednisolone as an adjuvant to local anesthetics

INTERVENTIONS:
Drug: TAPB with dexamethasone as an adjuvant to local anesthetics — patients will receive TAPB with dexamethasone as an adjuvant to bupivacaine and lidocaine local anesthetics
  Arms: Group TAPB-D (n=25)
Drug: TAPB with methylprednisolone as an adjuvant to local anesthetics — patients will receive TAPB with methylprednisolone as an adjuvant to bupivacaine and lidocaine local anesthetics
  Arms: Group TAPB-M (n=25)

SUMMARY:
The aim of this work to compare between the efficacy of ultrasound guided TAP block with dexamethasone as an adjuvant versus ultrasound guided TAPB with methyl prednisolone as an adjuvant to local anesthetic for postoperative pain management in lower abdominal hysterectomy procedures.

DETAILED DESCRIPTION:
Patients will be divided in to two groups; TAPB with dexamethasone as an adjuvant to local anesthetic Gr A(n=25) and TAPB with methyl prednisolone as an adjuvant to local anesthetic Gr B(n=25).

By the end of surgery and with the patient in supine position and after covering of surgery site, preparing the skin with povidone iodine, a high frequency (5-10 MHZ) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA) will be placed transversally on abdominal wall between lower costal margin and iliac crest near midline. After identifying the rectus abdominis muscle, we will gradually move the ultrasound probe laterally to identify the transversus abdominis muscle lying posterior to the rectus muscle. A 22 G echogenic needle using the in plane technique will be inserted medially aiming towards the iliac crest, then 30ml total volume of 0.25 plain bupivacaine 1.5mg/kg with lidocaine 1% 3mg/kg with 8mg dexamethasone in group A patients and 30ml total volume of 0.25 plain bupivacaine 1.5mg/kg with lidocaine 1% 3mg/kg with 50 mg methylprednisolone in group B patients.

Vital signs (H.R and non invasive blood pressure) will be recorded at the onset of the block then every 20 min for an hour then every 4hrs for 12 hrs. post operative

Postoperative:

Paracetamol every 8 hours and ketorolac every 12 hours should be given as a part of multimodal analgesia and nalbuphine given as rescue analgesia and included in secondary outcomes

Post-operative assessment and analgesic regimen

Post operative pain assessment using V.A.S will be assessed (0-10) (11) (as zero refer to no pain and 10 refer to the worst pain) after 1h of the block then every 4hrs for 12 hrs. then every 8hrs for 48 hrs then after 72hrs . The patient will be given Paracetamol every 8 hours and ketorolac every 12 hours The time to the first request of rescue post operative analgesic will be recorded, when the patient complain of pain (V.A.S> 3) intravenous nalbuphine 5mg will be given, total dose of nalbuphine will be recorded /24hrs.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II.
* Age 20-45 years.
* Undergoing lower abdominal hysterectomies.

Exclusion Criteria:

* Patient refusal
* Patients with coagulopathy.
* Hypertensive patients.
* Diabetic patients.
* Morbid obesity
* Allergy to the used drugs

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
postoperative pain score by Visual analogue score at 48 hrs. | 48 hours
  postoperative pain score by Visual analogue score at 48 hours Post operative pain assessment using Visual analogue score which is numerical score from (0-10) (zero refer to no pain and 10 refer to the worst pain)

SECONDARY OUTCOMES:
Time to first analgesic request of rescue analgesia | 24 hours
  Time to first analgesic request of nalbuphine as a rescue analgesia
Total consumption of Nalbuphine in 1st 24 hours | 24 hours
  Total consumption of Nalbuphine in 1st 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No